CLINICAL TRIAL: NCT01108224
Title: Psychosocial Group Intervention to Patients With Primary Breast Cancer - Psychosocial and Survival Outcome From a Randomised Study
Brief Title: Psychotherapy to Patients With Primary Breast Cancer - Psycho-social and Survival Outcome From a Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Responsible Party: Ellen H. Boesen, MSc, PhD, Danish Cancer Society
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Camma 2003
Record Dates: First submitted 2010-02-16; First posted 2010-04-21 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2004-01

CONDITIONS: Breast Cancer
Keywords: Quality of life; Coping; Social relations; Survival; Psychotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychiatric Rehabilitation; Patient Education as Topic; Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial support (Experimental)
  Interventions: Behavioral: Psychosocial support
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Psychosocial support — Psycho-social group intervention including patient-education for 6 h per week for 2 weeks and group therapy 2½ h for 8 weeks
  Other Names: Patient-education and group therapy
  Arms: Psychosocial support

SUMMARY:
The purpose of this study is to determine whether an intervention to breast cancer patients including psycho-education and group psychotherapy can enhance quality of life and survival.

DETAILED DESCRIPTION:
PURPOSE: This randomized study included patients diagnosed with breast cancer who participated in an intervention including education and group psychotherapy lasting 10 weeks after surgery. The purpose of the study was to enhance Quality of Life, coping and social relations and to support the women when going through treatment. PATIENTS AND METHODS: We randomly assigned 210 patients with primary breast cancer to a control or an intervention group. Patients in the intervention group were offered 2 weekly 6-hour sessions of psycho-education and eight weekly 2-hour sessions of group psychotherapy. Participants and nonparticipants were followed up for QoL, coping and social relations after one, six and twelve months post intervention and on vital status 5 years after surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were 18-70 years of age with stage I-IIIA primary breast cancer

Exclusion Criteria:

* Distant metastasis
* Not speaking or understanding Danish
* Over 71 years
* Other life-threatening diseases
* Brain-damaged

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 months post intervention
  Does Quality of Life enhance among a group of primary breast cancer patients who participate in a psychosocial group intervention compared to a control group of primary breast cancer patients who do not recieve any psychosocial intervention?

SECONDARY OUTCOMES:
Survival | 5 years post surgery
  Does primary breast cancer patients who participate in a psychosocial intervention survive for longer time compared to a control group of primary cancer patients who do not participate in any intervention?

CONTACTS AND LOCATIONS:
Overall Officials: Ellen H Boesen, MSc, Phd, Principal Investigator — Institute of Cancer Epidemiology, Danish Cancer Society, Strandboulevarden 49, DK-2100; Christoffer Johansen, DSc (Med), Study Chair — Institute of Cancer Epidemiology, Danish Cancer Society, Strandboulevarden 49, DK-2100